CLINICAL TRIAL: NCT04342975
Title: A Phase II, Randomized, Double-blinded, Placebo-controlled Clinical Trial to Evaluate the Efficacy of BASIS™ (Nicotinamide Riboside and Pterostilbene) Treatment for Kidney Protection in Patients Treated by Complex Aortic Aneurysm Repair and Aortic Arch Reconstruction
Brief Title: Protection From Acute Kidney Injury (AKI) With Basis™ Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Elysium Health (Industry)
Responsible Party: Principal Investigator, Bernardo C. Mendes, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-000162
Record Dates: First submitted 2019-08-13; First posted 2020-04-13 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: AKI
Keywords: AKI; open vascular surgery; endovascular surgery; aortic arch reconstruction; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — nicotinamide-beta-riboside; Pterocarpus marsupium; Radial Basis Function Networks

STUDY DESIGN:
Intervention Model Description: This study is a single-center, prospective, randomized, double-blinded, placebo-controlled phase II clinical trial to evaluate the efficacy of "NAD+ supplementation" with Basis™ (Nicotinamide Riboside and Pterostilbene) in preventing acute kidney injury (AKI) in patients undergoing complex aortic aneurysm repair and open aortic arch reconstruction.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Basis (Active Comparator): The investigational product, Basis™, contains a synthetic NR that is nature-identical to naturally-occurring NR, does not induce flushing or pruritus and has no effect on lipid levels. Also contains Pterostilbene (Ptero) that is a stilbenoid compound, characterized by two aromatic rings connected by a methylene bridge backbone, and it has two methoxy groups and one hydroxyl group extending from the aromatic rings.
  Interventions: Drug: Nicotinamide Riboside + Pterostilbene
- Placebo (Placebo Comparator): Correspondent placebo, a capsule not containing the active component.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicotinamide Riboside + Pterostilbene — It will be administered a total of 1000 mg/day of NR and 200 mg/day of Ptero in a regimen of 2 capsules of Basis™ (each capsule 250 mg of NR and 50 mg of Ptero) 2 times a day by mouth for 2 weeks before surgery and 6 weeks after surgery. Each intake has to be apart from each other by, at least, 6 hours of interval.
  Other Names: Basis
  Arms: Basis
Drug: Placebo — The correspondent placebo will be administered in a regimen of 2 capsules 2 times a day by mouth for 2 weeks before surgery and 6 weeks after surgery. Each intake has to be apart from each other by, at least, 6 hours of interval.
  Arms: Placebo

SUMMARY:
This study is a single-center, prospective, randomized, double-blinded, placebo-controlled phase II clinical trial to evaluate the efficacy of "NAD+ supplementation" with Basis™ (Nicotinamide Riboside and Pterostilbene) in preventing acute kidney injury (AKI) in patients undergoing complex aortic aneurysm repair and open aortic arch reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* A patient may be included in the study if the following conditions are present:

  1. Male or female;
  2. Age > 18 years old;
  3. Patients who match the criteria for indication of elective open aortic arch replacement or repair:

     1. Total arch;
     2. Non-total arch;
  4. Patients who match the criteria for indication of elective complex aortic aneurysm repair has to respect the following conditions:

     a. Patients undergoing complex aortic aneurysm open reconstruction with a suprarenal clamp; i. thoracoabdominal aortic aneurysms Crawford extent I to IV ; ii. abdominal aortic aneurysms of juxtarenal, pararenal, or paravisceral type; b. For endovascular approach: i. patients with pararenal or thoracoabdominal aortic aneurysms Crawford extent I to IV and known stage III or IV of chronic kidney disease (CKD); ii. patients with pararenal or thoracoabdominal aortic aneurysms Crawford extent I to IV and solitary or single functioning kidney and known stage III or IV CKD;
  5. Patients will be allowed to participate in concomitant endovascular aortic stent-graft trials and prospective cohort studies as long as these do not involve another investigational study drug.

Exclusion Criteria:

* Patients must be excluded from the study if any of the following conditions are true:

5.2.1 General Exclusion Criteria

1. Unwilling to comply with the follow-up schedule;
2. Inability or refusal to give informed consent by the patient or a legally authorized representative;
3. Pregnant or breastfeeding;
4. Subject who takes multivitamins containing vitamin B3 derivatives in a dose > 200 mg/day; 5.2.2 Clinical / Laboratory Exclusion Criteria
5. Renal failure defined as eGFR< 15 mL/min/1.73m2
6. Patients in permanent Renal Replacement Therapy;
7. Patients with chronic liver disease: Child-Pugh score class B and C; 5.2.3 Medication Exclusion Criteria
8. Patients in chemotherapy scheme;
9. Patients taking any immunosuppressant, except for corticosteroids;
10. Patients taking any of these well-known P-glycoprotein substrates: digoxin, fexofenadine, indinavir, sirolimus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
AKI | 6 months
  The primary endpoint will be change in incidence of AKI measured by estimated glomerular filtration rate (eGFR) using the RIFLE criteria.

SECONDARY OUTCOMES:
Myocardial infarction | 6 months
  The secondary endpoint will be change in the incidence of myocardial infarction
Bowel ischemia | 6 months
  The secondary endpoint will be change in the incidence of bowel ischemia
Spinal cord injury | 6 months
  The secondary endpoint will be change in the incidence of spinal cord injury
Nicotinamide Adenine Dinucleotide (NAD), Nicotinamide Mononucleotide (NMN), and Nicotinamide Riboside (NR) | 6 months
  NAD, NMN, NR levels in peripheral blood mononuclear cells (PBMCs)
Tissue Inhibitor of Metalloproteinases 2 (TIMP2), Kidney Injury Molecule 1 (KIM-1), Insulin-like Growth Factor-binding Protein 7 (IGFBP7) | 6 months
  TIMP2, KIM-1, IGFBP7 levels in urine
Quinolinate and Tryptophan | 6 months
  Quinolinate and Tryptophan levels in urine

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Mendes, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials